CLINICAL TRIAL: NCT03664830
Title: A Pilot Study To Evaluate The Safety And Feasibility of Hematopoietic Progenitor Cell Mobilization With Plerixafor as Part of a Gene Therapy Strategy in Sickle Cell Disease
Brief Title: Safety of Blood Stem Cell Mobilization With Plerixafor in Patients With Sickle Cell Disease
Acronym: PISMO
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17426
Record Dates: First submitted 2018-09-07; First posted 2018-09-11 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Sickle Cell Disease
Keywords: plerixafor; sickle cell disease; mobilization; hematopoietic stem cell; gene therapy
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — plerixafor

STUDY DESIGN:
Intervention Model Description: Each SCD research participant will receive up to two subcutaneous injections of plerixafor (starting dose level: 240 µg/kg/dose)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Plerixafor (Experimental): Up to two subcutaneous injections of plerixafor (starting dose level: 240 µg/kg/dose)
  Interventions: Drug: Plerixafor

INTERVENTIONS:
Drug: Plerixafor — Up to two subcutaneous injections of plerixafor (starting dose level: 240 µg/kg/dose)

SUMMARY:
The objective of this study is to investigate if up to two injections of plerixafor represent a safe and effective strategy to mobilize adequate numbers of CD34+ hematopoietic stem progenitor cells (HSPC) for autologous hematopoietic cell transplantation (HCT) in sickle cell disease (SCD) patients

DETAILED DESCRIPTION:
Allogeneic hematopoietic cell transplantation (HCT) is the only curative option for sickle cell disease (SCD) patients but its use is significantly limited by the lack of compatible donors. Gene therapy using autologous hematopoietic stem cell (HSC) transplantation represents an alternative approach but requires the collection of significant numbers of cells. Severe adverse events have been observed in SCD patients after mobilization using the standard agent granulocyte colony-stimulating factor (G-CSF), and bone marrow harvesting is also associated with side effects. The use of a single administration of plerixafor has been suggested as an alternative mobilization strategy in SCD but may not mobilize sufficient number of HSC. In this study, our primary objective is to assess if up to two injections of plerixafor (starting dose level: 240 µg/kg/dose) are safe in SCD patients and can recruit enough blood stem cells needed for future gene therapy.

ELIGIBILITY:
Inclusion Criteria:

* Weight between 50 and 120 kg;
* Karnofsky performance status (KPS) ≥70%;
* Confirmed diagnosis of sickle cell disease with βS/βS or βS/β0 or βS/β+ genotype;
* Must have had one or more of the following events in the 2 year period preceding enrollment:

  * History of ≥2 severe vaso-occlusive pain crises (VOC) (or at least two episodes in the year preceding the setting up of regular transfusion protocol). A severe VOC is defined as an episode of pain lasting more than 2 hours severe enough to require care at a medical facility.
  * History of ≥1 episodes of acute chest syndrome despite the institution of supportive care measures (i.e. asthma therapy and/or hydroxyurea)
  * Clinically significant neurological event (stroke) or any neurological deficit lasting 24 hours. A stroke is defined as a sudden neurological change lasting more than 24 hours that is accompanied by cerebral magnetic resonance imaging (MRI) changes.
  * Prior treatment with regular RBC transfusion therapy, defined as receiving ≥8 transfusions per year for >1 year to prevent vaso-occlusive clinical complications (i.e. pain, stroke, and acute chest syndrome)
  * Osteonecrosis of two or more joints;
  * Anti-erythrocyte alloimmunization (>2 antibodies);
  * Presence of sickle cell cardiomyopathy documented by Doppler echocardiography;
  * Presence of any significant cerebral abnormality such as stenosis or occlusions on magnetic resonance imaging (MRA)
* Meet current eligibility requirements for donation for mobilization at the COH DAC;
* Adequate renal function: defined as a creatinine estimated FDR (eGFR) of ≥60 ml/min;
* Adequate liver function: defined by a serum conjugated (direct) bilirubin <2.5x upper limit of normal (ULN) for age; AST and ALT <5x ULN for age as per laboratory;
* Adequate cardiac function: defined as left ventricular ejection fraction >50%;
* Adequate hematologic parameters: WBC ≥2.5 x 10^9/L; platelet count ≥120 x10^9/L; hemoglobin >8 g/dL;
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry.

Exclusion Criteria:

* Diagnosed with alpha thalassemia (two or more gene deletions or any α-globin structural variants);
* Seropositivity for HIV-1/2 (Human Immunodeficiency Virus) or HTLV-1/2(Human T-Lymphotropic Virus);
* Evidence of uncontrolled bacterial, viral, or fungal infections (currently taking medication and progression of clinical symptoms) within one month prior to treatment. Participants with fever should await resolution of symptoms before starting the treatment;
* Any clinically significant active infection which, in the opinion of the investigator, would require significant medical intervention;
* Abnormal pulmonary function tests (adults with mild or moderate obstruction or restriction or diffusion defects are eligible, per Investigator discretion).
* History of pulmonary hypertension, proven by cardiac catheterization;
* History of malignancy or immunodeficiency disorder, (i.e., subjects with prior malignancy must be disease-free for 5 years), except curatively-treated basal cell carcinoma or cutaneous squamous cell carcinoma;
* Participation in any study with an investigational agent or medical device within 90 days of screening;
* Major surgery in the past 30 days;
* Prior receipt of any gene transfer product;
* Bone marrow harvest in the past year;
* Known myelodysplasia of the bone marrow or abnormal bone marrow cytogenesis;
* Known hypersensitivity to plerixafor or any excipient contained in Mozobil;
* G-CSF or plerixafor medication within 4 weeks of treatment;
* Pregnant or nursing women;
* Any condition or chronic physical, neurological, or mental illness, which in the opinion of the investigator, makes participation ill advised.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2026-08-03 (Estimated); Study Completion 2026-08-03 (Estimated)

PRIMARY OUTCOMES:
Toxicities | 120 hours (5 days) from the last injection of plerixafor
  Scored using the Common Terminology Criteria for Adverse Events (CTCAE) of the National Cancer Institute (NCI) version 4.03

SECONDARY OUTCOMES:
Stem cell mobilization feasibility | 6 hours after the first injection of plerixafor.
  Assessed by measuring the number of mobilized CD34+ cells/µL of peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Leo Wang, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States